CLINICAL TRIAL: NCT01841489
Title: A Phase 1, Open-Label, Adaptive Study of Novel GS-9973 Tablet Formulations to Evaluate the Effect of Acid Reducing Agents, Relative Bioavailability, and Food Effect on GS-9973 Pharmacokinetics
Brief Title: A Phase 1 Study of Novel GS-9973 Tablet Formulations to Evaluate the Effect of Acid Reducing Agents, Relative Bioavailability, and Food Effect on GS-9973 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-339-0111
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental)
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment G; Drug: Treatment I
- Sequence 2 (Experimental)
  Interventions: Drug: Treatment A; Drug: Treatment C; Drug: Treatment H; Drug: Treatment J
- Sequence 3 (Experimental)
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment G; Drug: Treatment I
- Sequence 4 (Experimental)
  Interventions: Drug: Treatment D; Drug: Treatment F; Drug: Treatment H; Drug: Treatment J

INTERVENTIONS:
Drug: Treatment A — 1600 mg GS-9973 (Formulation 1)
  Arms: Sequence 1; Sequence 2
Drug: Treatment B — 1600 mg GS-9973 (Formulation 1) plus 20 mg omeprazole
  Arms: Sequence 1
Drug: Treatment C — 1600 mg GS-9973 (Formulation 1) plus 40 mg famotidine
  Arms: Sequence 2
Drug: Treatment D — 1600 mg GS-9973 (Formulation 2)
  Arms: Sequence 3; Sequence 4
Drug: Treatment E — 1600 mg GS-9973 (Formulation 2) plus 20 mg omeprazole
  Arms: Sequence 3
Drug: Treatment F — 1600 mg GS-9973 (Formulation 2) plus 40 mg famotidine
  Arms: Sequence 4
Drug: Treatment G — 1600 mg GS-9973 (Reference formulation)
  Arms: Sequence 1; Sequence 3
Drug: Treatment H — 1600 mg GS-9973 (Formulation 1 or Formulation 2, based on results from Part A)
  Arms: Sequence 2; Sequence 4
Drug: Treatment I — An alternate dose of the chosen formulation from Part A up to 1200 mg administered twice-daily
  Arms: Sequence 1; Sequence 3
Drug: Treatment J — An alternate dose of the chosen formulation from Part A up to 1200 mg administered twice-daily
  Arms: Sequence 2; Sequence 4

SUMMARY:
This is a Phase 1, Open-Label, Adaptive Study of Novel GS-9973 Tablet Formulations to Evaluate the Effect of Acid Reducing Agents, Relative Bioavailability, and Food Effect on GS-9973 Pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Must have a body mass index (BMI) range of approximately 19 to 30 kg/m2
* Must have a minimum weight of 45 kg
* Females of childbearing potential must have negative serum pregnancy tests at screening and baseline and must practice at least 1 reliable method of contraception as defined by the protocol

  * Female subjects who utilize hormonal contraceptive as 1 of their birth control methods must have used the same method for at least 3 months prior to study dosing
* Male subjects must agree to use condoms during heterosexual intercourse and avoid sperm donation from Day -1 until 90 days following the last dose of study medication
* Must refrain from blood donation throughout the study period
* Must, in the opinion of the Investigator, be in good general
* Must be a non- or light smoker, eg, less than 10 cigarettes per day

Exclusion Criteria:

* Pregnant or lactating subjects
* Use of prescribed or over-the-counter medications that affect gastric pH
* History of severe peptic ulcer disease, GERD, or other diseases requiring prolonged(>6 weeks) medication or surgical therapy to modify gastric pH
* Have a history of clinically significant cardiac abnormalities or presence of clinically significant abnormality on 12-lead ECG.
* Have a history of any cancer requiring systemic chemotherapy or radiation
* Have a history of bleeding disorders
* Have a history of liver disorders
* Current acute infection or history of acute infection within 7 days
* Have a recent history of alcohol or illicit drug abuse and/or have a positive test for selected drugs of abuse
* Have a positive hepatitis screen or positive Human Immunodeficiency Virus antibody test
* Have participated in another clinical trial within 28 days
* Have received transfusion of blood or plasma products within 6 months
* Have donated > 500 mL blood within 56 days
* Are unable or unwilling to comply with study restrictions, return for follow-up appointments, or other considerations, which in the opinion of the Investigator, would make the candidate unsuitable for study participation
* Current or historical medical condition that is deemed to be of medical significance by the Investigator
* Have used prescription medications, over the counter products, herbal remedies and nutritional supplements within 7 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for GS-9973 | Up to 3 months
  The primary outcome measure is the pharmacokinetic (PK) parameters for GS-9973 including AUC and Cmax.

SECONDARY OUTCOMES:
Secondary pharmacokinetic parameters for GS-9973 | Up to 3 months
  A secondary outcome measure is the pharmacokinetic parameters for GS-9973 including Ctau and AUClast.
Incidence of Adverse Events | Up to 3 months
  A secondary outcome measure is the safety and tolerability of GS-9973 which will be evaluated by the incidence of AEs including assessment of clinical laboratory test findings, physical examinations, 12-lead ECG abnormalities, and vital signs measurements.
Blood PD parameters for GS-9973 | Up to 3 months
  A secondary outcome measure is the blood pharmacodynamic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hawkins, MD, Study Director — Gilead Sciences
Locations (1):
- Investigational Site, Daytona Beach, Florida, United States